CLINICAL TRIAL: NCT05527314
Title: Effect of Total Intravenous Anesthesia With Remimazolam vs Sevoflurane Inhalation Anesthesia on Incidence of Emergence Agitation and Complications in Children Undergoing Ophthalmic Surgery
Brief Title: Effect of Remimazolam vs Sevoflurane Anesthesia on Incidence of Emergence Agitation and Complications in Children Undergoing Ophthalmic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-EA-1
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Emergence Agitation; Remimazolam; Sevoflurane; Pediatric Ophthalmic Surgery; Anesthesia, General
Keywords: Anesthesia, General; Pediatric ophthalmic surgery; Emergence Agitation; Remimazolam; Sevoflurane
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Sevoflurane; Fentanyl; cisatracurium; Remifentanil

STUDY DESIGN:
Intervention Model Description: This is a RCTs.
Who Masked: Participant, Outcomes Assessor
Masking Description: Care provider and investigator (anesthesiologist) cannot be blinded for different appearance of sevoflurane and remimazolam.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Experimental): 1. Induction of anesthesia Slowly inject Remimazolam 0.4-0.8 mg/kg (about 1 minute) until loss of consciousness (LoC), if the degree of sedation is insufficient, additional Remimazolam (0.05 mg/kg each time) is allowed. After the LoC, fentanyl 3-4 ug/kg and cisatracurium besilate 0.1 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  2. Maintenance of anesthesia Remimazolam 1~2 mg/kg/h and remifentanil 0.1~0.3 ug/kg/min are injected intravenously to maintain sedation and assistant analgesia, and cisatracurium besilate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 20 %.
  Interventions: Drug: Remimazolam; Drug: Fentanyl; Drug: Cisatracurium Besylate; Drug: Remifentanil
- Sevoflorane (Active Comparator): 1. Induction of anesthesia After the sevoflurane volatilization tank is adjusted to 8 % and the fresh gas flow rate is 5 L/min, the suitable mask connects with the outlet of the loop and covers the nose of the child. After the LoC, the sevoflurane volatilization tank is set to 3 % and the fresh gas flow rate is 2 L/min to maintain autonomous respiration. At the same time, fentanyl 3-4 ug/kg and cisatracurium besilate 0.1 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  2. Maintenance of anesthesia Continuous inhalation of sevoflurane concentration 2 %-3 % and remifentanil 0.1-0.3 ug/kg/min intravenous pump to maintain sedation and assistant analgesia, and cisatracurium besilate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 20 %.
  Interventions: Drug: Sevoflurane; Drug: Fentanyl; Drug: Cisatracurium Besylate; Drug: Remifentanil

INTERVENTIONS:
Drug: Remimazolam — Anesthesia was induced with Remimazolam 0.4-0.8 mg/kg (about 1 minute) by intravenous injection until the loss of consciousness (LoC), followed by remimazolam 1-2 mg/kg/h until the end of surgery.
  Arms: Remimazolam
Drug: Sevoflurane — Anesthesia was induced with 8 % Sevoflorane by sevoflurane volatilization tank until the loss of consciousness (LoC), followed by 2 %-3 % Sevoflorane until the end of surgery.
  Arms: Sevoflorane
Drug: Fentanyl — Anesthesia was induced with fentanyl 3-4 ug/kg by intravenous injection after the LoC.
Drug: Cisatracurium Besylate — Anesthesia was induced with cisatracurium besilate 0.1 mg/kg by intravenous injection after the LoC. And the cisatracurium besilate 0.02 mg/kg is allowed to add as appropriate during the operation.
Drug: Remifentanil — After the LoC, remifentanil 0.1~0.3 ug/kg/min inject intravenously until the end of surgery.

SUMMARY:
As a novel ultra-short-acting benzodiazepines drugs, Remimazolam has been accepted for induction and maintenance of clinical anesthesia. Compared to the traditional benzodiazepines drugs, Remimazolam combines the safety of midazolam with the effectiveness of propofol, and also has the advantages of acting quickly, short half-life, no injection pain, slight respiratory depression, independent of liver and kidney metabolism, long-term infusion without accumulation, and has a specific antagonist: flumazenil. This study aims to investigate whether Remimazolam reduces the incidence of emergence agitation in children after ophthalmic surgery, compared to sevoflurane (RCT).

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ-Ⅱ
2. Aged 3-8 years, weight > 10 kg, sex was not limited；
3. Children were scheduled for selective ophthalmic surgery under general anesthesia,

Exclusion Criteria:

1. Respiratory infection was present within 4 weeks before surgery.
2. Potential or presence of difficult airways, airway obstruction, sleep apnea, and other contraindications to general anesthesia.
3. The blood routine or blood biochemical indexes were obviously abnormal.
4. Allergy or hypersensitive reaction to test drug, including remimazolam, sevoflurane, and remifentanil.
5. Any child who has taken benzodiazepines in the last 3 months.
6. Unable to cooperate to complete the test, and the guardian refused to attend.
7. Other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence agitation | Duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 30 minutes
  The PAED scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20. The degree of emergence delirium increased directly with the total score. PAED scale >12 at any time indicates presence of emergence agitation.
The incidence of emergence agitation | Duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 30 minutes
  The Watcha scale consists of four items and scores >2 at any time indicates presence of emergence agitation.
The incidence of emergence agitation | Duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 30 minutes
  The 5-point scale consists of five items. The scores ≥4 and lasts for more than 5 minutes indicate presence of emergence agitation.

SECONDARY OUTCOMES:
Systolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  "30 minutes before induction", "immediately after intubation", "every 5 minutes after intubation until the child leaves the post-anesthesia care unit and returns to the ward".
Diastolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  "30 minutes before induction", "immediately after intubation", "every 5 minutes after intubation until the child leaves the post-anesthesia care unit and returns to the ward".
Mean pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  "30 minutes before induction", "immediately after intubation", "every 5 minutes after intubation until the child leaves the post-anesthesia care unit and returns to the ward".
Heart rate | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  "30 minutes before induction", "immediately after intubation", "every 5 minutes after intubation until the child leaves the post-anesthesia care unit and returns to the ward".
Recovery times | Up to 30 minutes after operation
  The period from discontinuation of anesthetic drugs to the recovery of the child's self-consciousness and can respond correctly to external stimuli.
Delayed emergence | Up to 30 minutes after operation
  Delayed emergence is defined as failure to shake hands and no significant response to nociceptive stimuli more than 30 minutes after surgery.
Postoperative Pain | During the recovery from anesthesia.
  The FLACC scale consists of fIve items. Each item is scored 0-2 yielding a total between 0 and 10. The degree of pain increased directly with the total score.
Complication | During the perioperative period
  All the perioperative complications are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang University, Nanchang, Jiangxi, China